CLINICAL TRIAL: NCT04727021
Title: Single-dose, Open-label, Randomized, 2-way Crossover Bioequivalence Study of 20 mg Granules for Oral Suspension Rivaroxaban Versus 20 mg Tablets Rivaroxaban Under Fed Condition in Healthy Subjects
Brief Title: A Trial to Learn How Much Rivaroxaban Gets Into the Blood When Taken in Different Forms and How Safe They Are in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19366; 2017-000609-18 (EudraCT Number)
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Rivaroxaban; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A: Single oral dose of a 20 mg tablet rivaroxaban (Experimental): 2-way crossover: The subjects will receive the following treatments in a randomized order:
  * Treatment A: Single oral dose of a 20 mg tablet rivaroxaban, administered under fed conditions
  * Treatment B: Single oral dose of 20 mg rivaroxaban, granules for oral suspension administered under fed conditions.
  Interventions: Drug: 20 mg tablet rivaroxaban
- Treatment B: Single oral dose of 20 mg rivaroxaban, granules (Experimental): 2-way crossover: The subjects will receive the following treatments in a randomized order:
  * Treatment A: Single oral dose of a 20 mg tablet rivaroxaban, administered under fed conditions
  * Treatment B: Single oral dose of 20 mg rivaroxaban, granules for oral suspension administered under fed conditions.
  Interventions: Drug: 20 mg rivaroxaban, granules for oral suspension

INTERVENTIONS:
Drug: 20 mg tablet rivaroxaban — Single oral dose of a 20 mg tablet rivaroxaban, administered under fed conditions
  Arms: Treatment A: Single oral dose of a 20 mg tablet rivaroxaban
Drug: 20 mg rivaroxaban, granules for oral suspension — Single oral dose of 20 mg rivaroxaban, granules for oral suspension administered under fed conditions.
  Arms: Treatment B: Single oral dose of 20 mg rivaroxaban, granules

SUMMARY:
Researchers are looking for a better way to treat venous thromboembolic disease, also known as VTE. In people with VTE, blood clots form in the veins of the legs, groin, or arms. These clots or a piece of a clot can break free and move around the body in the blood vessels. These clots can block small blood vessels, causing other conditions like high blood pressure, heart attack, and stroke.

Before people with a medical condition can take an approved treatment in a new form, researchers do trials in healthy participants. This helps them understand how the new form acts in the body and to better understand its safety.

In this trial, the researchers will compare how much of the trial treatment gets into the blood when taken in 2 different forms in a small number of participants. The trial will include about 30 men who are aged 18 to 55.

In this trial, there will be 2 groups of participants. The participants will take rivaroxaban in the current tablet form and in a new liquid form 1 time. This was a "crossover" trial. In a crossover trial, all the participants will take both forms of the treatments, but in a different order.

During the trial, the participants will stay at their trial site 2 times for 5 days. But, the participants can be in the trial for up to about 6 weeks. During the trial, the doctors will take blood and urine samples and check the participants' heart health using an electrocardiogram (ECG) and measure the blood pressure. The participants will also answer questions about how they are feeling, if they have any medical problems, and about any medications they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects.
* Age: 18 to 55 years (inclusive) at the screening examination/visit.
* Race: White (Note: Clinical Data Interchange Standards Consortium definition of White: Denotes a person with European, Middle Eastern, or North African ancestral origin who identifies, or is identified, as White (Food and Drug Administration [FDA]).
* Body mass index (BMI): above/equal 18 and below/equal 29.9 kg/m2.
* Ability to understand and follow instructions.

Exclusion Criteria:

* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known or suspected liver disorders and bile secretion/flow
* Subjects with thyroid disorders as evidenced by assessment of thyroid stimulating hormone (TSH) levels outside the normal reference range at screening
* Personal or familial history of genetically muscular diseases
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies e.g. allergies to more than 3 allergens, allergies affecting the lower respiratory tract- allergic asthma, allergies requiring therapy with corticosteroids, urticaria) or significant non-allergic drug reactions
* Known disorders with increased bleeding risk (e.g., periodontosis, hemorrhoids, acute gastritis, peptic ulcer)
* Known sensitivity to common causes of bleeding (e.g. nasal)
* Clinically relevant findings in the electrocardiogram (ECG) such as a second- or third-degree atrioventricular (AV) block, prolongation of the QRS (QRS interval in ECG) complex over 120 msec or of the QTc-interval over 450 msec at the first screening visit
* Presence or history of arrhythmic disturbances; or known congenital QT (QT interval in ECG) prolongation
* Systolic blood pressure below 100 or above 140 mmHg
* Diastolic blood pressure below 50 or above 90 mmHg
* Heart rate below 50 or above 90 beats/ min

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
AUC of rivaroxaban granules for oral suspension vs. rivaroxaban tablet | From pre-dose up to 72 hours after drug administration
  AUC = area under the concentration vs. time curve from zero to infinity after single (first) dose
  Rivaroxaban Blood sampling for rivaroxaban pharmacokinetics in plasma.
AUC(0-tlast) of rivaroxaban granules for oral suspension vs. rivaroxaban tablet | From pre-dose up to 72 hours after drug administration
  AUC(0-tlast) = AUC from time 0 to the last data point > lower limit of quantification (LLOQ)
  Rivaroxaban Blood sampling for rivaroxaban pharmacokinetics in plasma.
Cmax of rivaroxaban granules for oral suspension vs. rivaroxaban tablet | From pre-dose up to 72 hours after drug administration.
  Cmax = maximum observed drug concentration in measured matrix after single dose administration
  Rivaroxaban Blood sampling for rivaroxaban pharmacokinetics in plasma.

SECONDARY OUTCOMES:
Number of treatment-emergent adverse events | Up to 7-14 days after the last administration
  Adverse events occurring in the period between the signing of the informed consent and the end of the follow-up phase.

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Mönchengladbach GmbH, Mönchengladbach, North Rhine-Westphalia, Germany